CLINICAL TRIAL: NCT03944915
Title: A Phase II Trial of Carboplatin, Paclitaxel, and Nivolumab Induction Therapy Followed by Response-stratified Locoregional Therapy for Patients With Locally Advanced, HPV-negative Head and Neck Cancer. The DEPEND Trial.
Brief Title: De-Escalation Therapy for Human Papillomavirus Negative Disease
Acronym: DEPEND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-0162
Record Dates: First submitted 2019-05-01; First posted 2019-05-10 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Human Papilloma Virus; Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Head and Neck; HPV-Related Squamous Cell Carcinoma; HNSCC
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Paclitaxel; Nivolumab; Radiation; Hydroxyurea; Fluorouracil; Filgrastim; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Chemotherapy (Experimental): Induction Therapy
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Nivolumab
- De-escalated Chemotherapy (Experimental): Radiation therapy with chemotherapy
  Interventions: Drug: Paclitaxel; Radiation: Radiation; Drug: Hydroxyurea Pill; Drug: 5-fluorouracil; Drug: Filgrastim Injection; Drug: Cisplatin

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be given through IV infusions for 30-60 minutes on day 1 of each cycle. Each cycle will last 21 days. There will be 3 cycles.
  Arms: Standard Chemotherapy
Drug: Paclitaxel — During Induction Therapy Paclitaxel (100 mg) will be given through IV infusions on days 1, 8 and 15 of each 21 day cycle. There will be 3 cycles.
  During Radiotherapy, paclitaxel will be given after a dose of radiation by IV infusion for 60 minutes after day 1 of radiotherapy.
Drug: Nivolumab — Nivolumab will be given through IV infusions at 360 mg on day 1 every 21 days for 3 cycles.
  Arms: Standard Chemotherapy
Radiation: Radiation — Patients will receive 4.5-5 cycles of radiation depending on response. Those with a positive response will receive radiation for 4.5 cycles with a total radiation dose of 66 Gy. Patients with a moderate or no response will receive 5 cycles with a total radiation dose of 70-75 Gy. 2 times a day for days 1-5 followed by a rest period for days 6-13
  Arms: De-escalated Chemotherapy
Drug: Hydroxyurea Pill — One dose of hydroxyurea pill by mouth at start of 5-FU infusion during radiotherapy cycle
  Arms: De-escalated Chemotherapy
Drug: 5-fluorouracil — 5-FU will be given by IV infusion continuously for 5 days during radiotherapy cycles
  Other Names: 5-FU
  Arms: De-escalated Chemotherapy
Drug: Filgrastim Injection — Filgrastim shot will be given if patient has certain side effects during radiotherapy cycle on days 6-12.
  Other Names: Filgrastim shot
  Arms: De-escalated Chemotherapy
Drug: Cisplatin — Radiotherapy may also be given with a different chemotherapy agent called cisplatin. This is the traditional standard of care chemotherapy regimen. In this case, the radiotherapy will be given once daily for 5 days per week. Cisplatin will be administered via IV once every 21 days for 2 or 3 cycles.
  Arms: De-escalated Chemotherapy

SUMMARY:
This study is looking to see if nivolumab, an immunotherapy drug, given with carboplatin and paclitaxel (2 chemotherapy agents) during induction therapy in advanced stage HPV negative patients can significantly shrink the subject's cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically confirmed locally advanced, non-metastatic, HPV-negative head and neck squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, nasopharynx, larynx, or sinuses.
2. Stage IV disease with the exception of nasopharyngeal tumor-3, node-2 (stage III) based of American Joint Committee on Cancer staging 8th edition
3. If a primary oropharyngeal squamous cell carcinoma is diagnosed, HPV must be ruled out by immunohistochemistry.
4. Availability of ≥10 unstained 5 micron slides. Patients who cannot fulfill this requirement will need to undergo a new biopsy prior to enrollment on study.
5. Patients must be at least 18 years of age.
6. Measurable disease (either primary site and/or nodal disease) by RECIST criteria.
7. No previous radiation or chemotherapy for a head and neck cancer.
8. No complete surgical resection for a head and neck cancer within 8 weeks of enrollment (although lymph node biopsy including excision of an individual node with presence of residual nodal disease, or surgical biopsy/excision of the tumor with residual measurable disease is acceptable.) No surgical procedures or biopsies will occur after baseline scans are performed and measurable lesions are identified.
9. Eastern Cooperative Oncology Group performance status 0-1
10. Normal Organ Function

    1. Leukocytes ≥ 3000/mm3
    2. Platelets ≥ 100,000/mm3
    3. Absolute neutrophil count ≥ 1,500
    4. Hemoglobin ≥ 9.0 gm/dL
    5. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5x upper limit of normal
    6. Alkaline phosphatase ≤ 2.5x upper limit of normal
    7. Albumin > 2.9 gm/dL
    8. Total bilirubin ≤ 1.5 mg/dL
    9. Creatinine clearance > 45 mL/min, normal within 2 weeks prior to start of treatment (Of note, the standard Cockcroft and Gault formula must be used to calculate creatinine clearance (CrCl) for enrollment or dosing)
11. Patients must sign a study-specific informed consent form prior to study entry. Patients should have the ability to understand and the willingness to sign a written informed consent document.
12. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug
13. Women must not be breastfeeding
14. Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 6 months after completing chemoradiation or receiving the last dose of consolidative nivolumab, whichever occurs latest.
15. Men who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 6 months after completing chemoradiation or receiving the last dose of consolidative nivolumab, whichever occurs latest.

Exclusion Criteria:

1. Unequivocal demonstration of distant metastatic disease (M1 disease).
2. Unidentifiable primary site.
3. Inter-current medical illnesses which would impair patient tolerance to therapy or limit survival. This includes but is not limited to ongoing or active infection, immunodeficiency, symptomatic congestive heart failure, pulmonary dysfunction, cardiomyopathy, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance. Patients with clinically stable and/or chronically managed medical illnesses that are not symptomatic and/or are not expected to impact treatment on protocol are still eligible (conditions to be reviewed by the PI to confirm eligibility)
4. Prior surgical therapy other than incisional/excisional biopsy or organ-sparing procedures such as debulking of airway-compromising tumors. Residual measurable tumor is required for enrollment as discussed above.
5. Patients receiving other investigational agents.
6. Diagnosis of immunodeficiency or is receiving systemic steroid therapy in excess of physiologic dose or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
7. Known history of active tuberculosis (Bacillus Tuberculosis infection).
8. Hypersensitivity to nivolumab or any other drug used in this protocol.
9. Prior systemic anti-cancer treatment within the last 8 weeks.
10. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or any tumors that are not likely to influence life expectancy in the subsequent 3 years without active treatment.
11. Has active autoimmune disease that has required systemic therapy in the past year (i.e. with steroids or immunosuppressive drugs). Replacement therapy e.g. levothyroxine, insulin, or physiologic corticosteroid doses for adrenal or pituitary insufficiency, etc. are not considered a form of systemic treatment.
12. Has known history of, or any evidence of active, non-infectious pneumonitis.
13. Has a history of HIV.
14. Has known active Hepatitis B or hepatitis C. If eradicated, patient is eligible.
15. Has received a live vaccine within 28 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, MD, Principal Investigator — University of Chicago
Locations (1):
- University Of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Rosenberg AJ, Juloori A, Jelinek MJ, Agrawal N, Cursio JF, Cipriani N, Lingen MW, Izumchenko E, Katipally R, Chin J, Ginat D, Pasternak-Wise O, Gooi Z, Blair E, Pearson AT, Haraf DJ, Vokes EE. Neoadjuvant Nivolumab Plus Chemotherapy Followed by Response-Stratified Chemoradiation Therapy in HPV-Negative Head and Neck Cancer: The DEPEND Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2025 May 1;11(5):492-501. doi: 10.1001/jamaoncol.2025.0081. PMID 40048190

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Chemotherapy: Induction Therapy
  Carboplatin: Carboplatin will be given through IV infusions for 30-60 minutes on day 1 of each cycle. Each cycle will last 21 days. There will be 3 cycles.
  Paclitaxel: During Induction Therapy Paclitaxel (100 mg) will be given through IV infusions on days 1, 8 and 15 of each 21 day cycle. There will be 3 cycles.
  During Radiotherapy, paclitaxel will be given after a dose of radiation by IV infusion for 60 minutes after day 1 of radiotherapy.
  Nivolumab: Nivolumab will be given through IV infusions at 360 mg on day 1 every 21 days for 3 cycles.
- De-escalated Chemotherapy: Radiation therapy with chemotherapy
  Paclitaxel: During Induction Therapy Paclitaxel (100 mg) will be given through IV infusions on days 1, 8 and 15 of each 21 day cycle. There will be 3 cycles.
  During Radiotherapy, paclitaxel will be given after a dose of radiation by IV infusion for 60 minutes after day 1 of radiotherapy.
  Radiation: Patients will receive 4.5-5 cycles of radiation depending on response. Those with a positive response will receive radiation for 4.5 cycles with a total radiation dose of 66 Gy. Patients with a moderate or no response will receive 5 cycles with a total radiation dose of 70-75 Gy. 2 times a day for days 1-5 followed by a rest period for days 6-13
  Hydroxyurea Pill: One dose of hydroxyurea pill by mouth at start of 5-FU infusion during radiotherapy cycle
  5-fluorouracil: 5-FU will be given by IV infusion continuously for 5 days during radiotherapy cycles
  Filgrastim Injection: Filgrastim shot will be given if patient has certain side effects during radiotherapy cycle on days 6-12.
  Cisplatin: Radiotherapy may also be given with a different chemotherapy agent called cisplatin. This is the traditional standard of care chemotherapy regimen. In this case, the radiotherapy will be given once daily for 5 days per week. Cisplatin will be administered via IV once every 21 days for 2 or 3 cycles.
Period: Overall Study
Arm/Group | Standard Chemotherapy | De-escalated Chemotherapy
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Chemotherapy: Standard chemoradiotherapy with paclitaxel, 5-FU, hydroxyurea and hyperfractionated, accelerated radiotherapy to 75 Gy encompassing GTV of primary and nodal disease as well as elective prophylactic nodal irradiation. OR Standard chemoradiotherapy with cisplatin and radiotherapy to 70 Gy encompassing GTV of primary and nodal disease as well as elective prophylactic nodal irradiation
- De-escalated Chemotherapy: De-escalated chemoradiotherapy with paclitaxel, 5-FU, hydroxyurea and hyperfractionated, accelerated radiotherapy to 66 Gy encompassing GTV of primary and nodal disease without elective prophylactic nodal irradiation. OR De-escalated chemoradiotherapy with cisplatin and radiotherapy to 66 Gy encompassing GTV of primary and nodal disease without elective prophylactic nodal irradiation.
- Total: Total of all reporting groups
Arm/Group | Standard Chemotherapy | De-escalated Chemotherapy | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 5 | 8 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (11.9) | 60.1 (12.4) | 58.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 19 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 16 | 19 | 35

OUTCOME MEASURES:

1. Primary Outcome: Deep Response Rate (DRR)
Description: DRR is 50% or greater response to induction therapy based on RECIST criteria. The objective is to intensify induction chemotherapy with the addition of an immune checkpoint inhibitor aimed at increasing the proportion of patients achieving a deep tumor response in order to subsequently allow risk-adapted definitive chemoradiotherapy in advanced stage HPV negative head and neck squamous cell cancer patients.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Chemotherapy | De-escalated Chemotherapy
Number analyzed (Participants) | 16 | 19
Participants | 16 | 19

2. Secondary Outcome: Progression Free Survival Rate (PFS)
Description: Progression free survival at 24 months after completing chemoradiation. PFS will be defined as the time from registration to the date of the first documented disease progression, clinical progression, or death due to any cause, whichever occurs first.
Time Frame: 26 months
Measure: Number (95% Confidence Interval); unit: percentage of patients in each arm
Arm/Group | Standard Chemotherapy | De-escalated Chemotherapy
Number analyzed (Participants) | 16 | 19
percentage of patients in each arm | 69 [40 to 86] | 69 [39 to 87]

3. Secondary Outcome: Overall Survival Rate (OS)
Description: Overall survival will be defined as the time between the date of registration and the date of death.
Time Frame: 26 months
Measure: Number (95% Confidence Interval); unit: percentage of patients in each arm
Arm/Group | Standard Chemotherapy | De-escalated Chemotherapy
Number analyzed (Participants) | 16 | 19
percentage of patients in each arm | 79 [47 to 93] | 74 [41 to 90]

4. Secondary Outcome: Locoregional Control After Completing Chemoradiation
Description: Assess disease control in all patients receiving induction chemoimmunotherapy and compare disease control between radiation arms.
Time Frame: 26 months
Measure: Number (95% Confidence Interval); unit: percentage of patients in each arm
Arm/Group | Standard Chemotherapy | De-escalated Chemotherapy
Number analyzed (Participants) | 16 | 19
percentage of patients in each arm | 93 [61 to 99] | 89 [63 to 97]

5. Secondary Outcome: Distant Control After Completing Chemoradiation
Description: Distant control will be defined as the percent of patients with disease progression below the clavicles. Comparison between the two radiation arms will be made.
Time Frame: 26 months
Measure: Number (95% Confidence Interval); unit: percentage of patients in each arm
Arm/Group | Standard Chemotherapy | De-escalated Chemotherapy
Number analyzed (Participants) | 16 | 19
percentage of patients in each arm | 90 [47 to 99] | 94 [63 to 99]

6. Other Pre Specified Outcome: Acute and Late Toxicity During Treatment
Description: Assess long term and late toxicities in all patients receiving induction therapy and risk-adapted chemoradiotherapy after deep response to induction therapy. Acute and late toxicities will be defined using the National Cancer Institute Common Terminology Criteria for Adverse Events. Comparisons will be made using Fisher's exact test. Acute and late toxicity during treatment and at 1 month, 3 months and 1 year post chemoradiation
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Chemotherapy | De-escalated Chemotherapy
Number analyzed (Participants) | 16 | 19
Participants | 0 | 0

7. Other Pre Specified Outcome: Enteral Tube Dependency
Description: Enteral tube dependency will be defined as continued necessity of any nutrition through enteral tube to maintain weight. The rate of enteral tube dependency will be described within the safety population and among each radiation treatment. Comparisons will be made using Fisher's exact test.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Standard Chemotherapy | De-escalated Chemotherapy
Number analyzed (Participants) | 16 | 19
participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 26 months
Arm/Group | Standard Chemotherapy | De-escalated Chemotherapy
All-Cause Mortality (participants affected / at risk) | 3/16 | 2/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 15/16 | 15/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Chemotherapy (N=16) | De-escalated Chemotherapy (N=19)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 6 (12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 3 (6) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 7 (7) | 7 (8)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 8 (8) | 7 (8)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 10 (11) | 7 (9)
Dysphagia (Gastrointestinal disorders) | 5 (6) | 5 (6)
Esophagitis (Gastrointestinal disorders) | 3 (4) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 15 (36) | 14 (34)
Nausea (Gastrointestinal disorders) | 7 (9) | 6 (8)
Oral pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (8) | 2 (4)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 9 (15) | 11 (25)
Chills (General disorders) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 3 (5) | 1 (1)
Fatigue (General disorders) | 3 (3) | 6 (7)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 2 (2) | 1 (1)
Paronychia (Infections and infestations) | 1 (2) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 14 (33) | 13 (25)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (7) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (2)
Weight loss (Investigations) | 4 (4) | 3 (3)
White blood cell decreased (Investigations) | 0 (0) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 5 (7) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 6 (9) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (7) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 10 (13) | 8 (11)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (8) | 4 (6)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (5) | 1 (1)
Delirium (Psychiatric disorders) | 1 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 4 (5)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 8 (9)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 7 (11) | 4 (6)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (10) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT03944915/Prot_SAP_000.pdf